CLINICAL TRIAL: NCT05586334
Title: Development and Clinical Evaluation of an Innovative Medical Device to Predict Preterm Birth: From Basic Research to Obstetric Emergencies
Brief Title: Development and Clinical Evaluation of an Innovative Medical Device to Predict Preterm Birth (PrediMAP)
Acronym: PrediMAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: APHP220187; 2022-A00588-35 (Other: ID-RCB Number)
Record Dates: First submitted 2022-07-28; First posted 2022-10-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Preterm Labor
Keywords: obstetrics; medical device; preterm labor; preterm birth; prediction
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: lack of result reporting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Collection of vaginal secretions — In all women included: Vaginal secretion sampling at the time of the obstetrical emergency consultation.
Biological: Collection of the placenta and the membranes — In cohort 1, for 30 patients at the Port Royal Maternity Hospital, the placenta and membranes will be collected after delivery
Other: Administration of EPDS questionnaire — In cohort 3, the EPDS questionnaire will be administered to all participants after the consultation in the emergency department.

SUMMARY:
The purpose of this study is to clinically validate the predictive performance (sensitivity and specificity) of the PrediMAP in-vitro diagnostic medical device to predict delivery within 7 days in the target population of women consulting obstetric emergencies for preterm labor (PTL).

DETAILED DESCRIPTION:
Preterm delivery (birth before 37 weeks of gestation) accounts for 12% of worldwide births each year: 15 million children. It is the leading cause of infant mortality. In France, it accounts for 60,000 births per year, 10,000 of them very preterm (before 32 weeks) and at very high risk of neonatal complications and childhood sequelae Given the high risks of death and of neurodevelopmental disabilities and learning disorders among survivors, preterm birth (PTB) is a major public health problem .

Over the past 30 years, measures to prevent preterm deliveries have not proved effective, and the incidence of PTB is rising or at best stable in most developed countries, including France. Important advances have nonetheless improved the management of pregnancies at risk of PTB and of preterm children.

From 100,000 to 150,000 women a year come to maternity unit EDs for symptoms suggesting PTL. Although fewer than half will be admitted to the hospital, our team has shown that PTL is the leading reason for hospitalization among pregnant women (45,000 admissions/year) in France [4]. In the USA, PTL is also the main cause of hospitalization during pregnancy, with costs estimated at $820 million annually . This hospitalization benefits only those women who finally do give birth preterm.

The PrediMAP project's ambition is to use new markers involved in the mechanism of PTL in clinical practice - biomarkers that are the fruit of more than 10 years of basic research at the Institut Cochin. The objective is to combine their measurement with clinical and ultrasound data to construct an algorithm to predict PTB within 7 days after the test, one that medical teams can use in obstetric EDs.

The final objective is to obtain a personalized prediction of delivery within 7 days via an algorithm integrated in the IVD-MD that includes clinical and ultrasound data with these biomarker measurements.

This study is conducted in 3 phases (3 cohorts).

* Objectives of Cohort 1 (Development) :

  1. Collect vaginal samples for development of the device
  2. Collect clinical and ultrasound data for the predictive algorithm
  3. Collect placenta and membrane samples to identify additional biomarkers
* Objective of Cohort 2 (Technical validation ): Validate technically the ergonomics and reliability of the bedside device
* Objective of Cohort 3 (Clinical performance) : Validate the clinical performance of the PrediMAP solution in the target population

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with live fetus(es)
* Emergency room visit between 22 and 34 days of pregnancy + 6 days
* For a suspicion of PTL defined by :

  * Uterine contractions (UC) objectified during the consultation (questioning, clinical examination, external tocography),
  * And/or clinical or ultrasound changes of the uterine cervix;
* OR for any other reason but with EC and/or clinical or ultrasound changes of the cervix on clinical examination
* Social security coverage or AME: patients receiving AME are at higher risk of PAD and preterm delivery.
* Signature of consent

Exclusion Criteria

* Age < 18 years;
* Premature rupture of membranes
* Patient in labor with imminent delivery.
* Total absence of social care
* Minor or protected adult (guardianship or curatorship)
* Persons who do not speak French and not accompanied by a French-speaking third party
* Multiple pregnancy >= 3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Delivery occurence 7 days after inclusion | Cohort 1 : assessed 15-21 days after inclusion of each patient. Cohort 3: assessed after end of follow-up (5.5 months).

SECONDARY OUTCOMES:
delivery occurrence 14 days after consultation | assessed after end of follow-up (5.5 months)
delivery <32 weeks of gestation, <34 weeks and <37 weeks | assessed after end of follow-up (5.5 months)
  Gestational age at delivery, in 4 categories.
neonatal mortality; | assessed after end of follow-up (5.5 months)
severe neonatal morbidity | assessed after end of follow-up (5.5 months)
  Defined by one or more of the following :
  * Bronchopumonary dyplasia
  * Necrotizing enterocolitis stage 2 or 3
  * Intraventricular haemorrhage stage 3-4
  * Periventricular leukomalacia
  * Retinopathy of prematurity stage >3
EPDS score at inclusion and after delivery | assessed after end of follow-up (5.5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne SIBIUDE, MD, PhD, Principal Investigator — APHP; François GOFFINET, Pr, Study Chair — APHP
Locations (1):
- Louis Mourier Hospital, Colombes, France

IPD SHARING:
Plan to Share IPD: No